CLINICAL TRIAL: NCT00105196
Title: A Study of Aripiprazole in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CN138-165
Record Dates: First submitted 2005-03-09; First posted 2005-03-10 (Estimated); Results first posted 2009-05-18 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2011-04

CONDITIONS: Major Depressive Disorder
Keywords: Single or recurrent; non-psychotic episode of Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Aripiprazole+ ADT
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo+ ADT

INTERVENTIONS:
Drug: Aripiprazole+ ADT — Tablets, Oral, 2 - 20 mg variable dose once daily, 14 weeks
  Other Names: Abilify
  Arms: A1
Drug: Placebo+ ADT — Tablets, Oral, 2 - 20 mg variable dose once daily, 14 weeks
  Arms: A2

SUMMARY:
The purpose of this 14 week, randomized, double-blind, placebo controlled study is to assess the safety and efficacy of aripiprazole to placebo as adjunctive treatment to an assigned open-label marketed antidepressant therapy (ADT) in patients with Major Depressive Disorder who demonstrate an incomplete response to a prospective eight week trial of the same assigned open-label marketed antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old who have experienced single or recurrent, non-psychotic episodes of Major Depressive Disorder, with the current episode of minimally 8 weeks in duration.
* Treatment history of an inadequate response to at least one and no more than three adequate antidepressant trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- United States (34):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Sharp Mesa Vista Hospital, San Diego, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Cns Clinical Research Group, Coral Springs, Florida
  - Medical College Of Georgia, Augusta, Georgia
  - Carman Research, Smyrna, Georgia
  - Uptown Research Institute, Llc, Chicago, Illinois
  - Cunningham Clinical Research, Llc, Edwardsville, Illinois
  - Comprehensive Neuroscience, Inc., Hoffman Estates, Illinois
  - Vine Street Clinical Research Center, Springfield, Illinois
  - Clinical Research Institute, Witchita, Kansas
  - Lsu Health Sciences Center, New Orleans, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Summit Research Network, Farmington Hills, Michigan
  - Summit Research Network, Flint, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Radiant Research Las Vegas, Las Vegas, Nevada
  - Behavioral Health Center, Charlotte, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Phebe Tucker, Md, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Southeast Health Consultants, Charleston, South Carolina
  - Usc School Of Medicine, Columbia, South Carolina
  - Community Clinical Research, Inc., Austin, Texas
  - Radiant Research, Slc, Salt Lake City, Utah
  - University Of Utah School Of Medicine, Salt Lake City, Utah
  - University Of Virginia, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin

REFERENCES:
- [Background] Berman RM, Fava M, Thase ME, Trivedi MH, Swanink R, McQuade RD, Carson WH, Adson D, Taylor L, Hazel J, Marcus RN. Aripiprazole augmentation in major depressive disorder: a double-blind, placebo-controlled study in patients with inadequate response to antidepressants. CNS Spectr. 2009 Apr;14(4):197-206. doi: 10.1017/s1092852900020216. PMID 19407731
- [Derived] Stewart TD, Hatch A, Largay K, Sheehan JJ, Marler SV, Berman RM, Nelson JC. Effect of symptom severity on efficacy and safety of aripiprazole adjunctive to antidepressant monotherapy in major depressive disorder: a pooled analysis. J Affect Disord. 2014 Jun;162:20-5. doi: 10.1016/j.jad.2014.03.017. Epub 2014 Mar 24. PMID 24766999
- [Derived] Fabian TJ, Cain ZJ, Ammerman D, Eudicone JM, Tang Y, Rollin LM, Forbes RA, Berman RM, Baker RA. Improvement in functional outcomes with adjunctive aripiprazole versus placebo in major depressive disorder: a pooled post hoc analysis of 3 short-term studies. Prim Care Companion CNS Disord. 2012;14(6):PCC.12m01394. doi: 10.4088/PCC.12m01394. Epub 2012 Dec 20. PMID 23585999
- [Derived] Dunner DL, Laubmeier KK, Manos G, Forbes RA, Baker RA, Berman RM. Beneficial effects of adjunctive aripiprazole in major depressive disorder are not dependent on antidepressant therapy history: a post hoc analysis of 3 randomized, double-blind, placebo-controlled trials. Prim Care Companion CNS Disord. 2012;14(6):PCC.12m01380. doi: 10.4088/PCC.12m01380. Epub 2012 Nov 22. PMID 23585997
- [Derived] Casey DE, Laubmeier KK, Marler SV, Forbes RA, Baker RA. Efficacy of adjunctive aripiprazole in major depressive disorder: a pooled response quartile analysis and the predictive value of week 2 early response. Prim Care Companion CNS Disord. 2012;14(3):PCC.11m01251. doi: 10.4088/PCC.11m01251. Epub 2012 May 31. PMID 23106023
- [Derived] Fava M, Dording CM, Baker RA, Mankoski R, Tran QV, Forbes RA, Eudicone JM, Owen R, Berman RM. Effects of adjunctive aripiprazole on sexual functioning in patients with major depressive disorder and an inadequate response to standard antidepressant monotherapy: a post hoc analysis of 3 randomized, double-blind, placebo-controlled studies. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m00994. doi: 10.4088/PCC.10m00994gre. PMID 21731833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After initial screening period (7-28 days), subjects enrolled into an 8-wk prospective treatment phase (single-blind placebo plus an investigator-assigned, open-label, marketed antidepressant therapy [ADT]). Patients who met criteria for incomplete response at the end of this phase were randomized into the 6-wk double-blind phase in a 1:1 ratio.
Groups:
- Aripiprazole + ADT: Subjects with a recorded baseline value at Week 8 and at least one recorded value on randomized study drug (aripiprazole). Missing baseline values were not imputed. Missing values on study drug were imputed using LOCF. Baseline values were not carried forward.
- Placebo + ADT: Subjects with a recorded baseline value at Week 8 and at least one recorded value on randomized study drug (placebo). Missing baseline values were not imputed. Missing values on study drug were imputed using LOCF. Baseline values were not carried forward.
Period: Overall Study
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Started | 177 | 172
Completed | 147 | 149
Not Completed | 30 | 23
Not completed — Lack of Efficacy | 2 | 3
Not completed — Adverse Event | 11 | 3
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Poor/noncompliance | 3 | 4
Not completed — Protocol Violation | 5 | 2
Not completed — pending surgery | 0 | 1
Not completed — marijuana use | 0 | 1
Not completed — Subject became unblinded | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole + ADT | Placebo + ADT | Total
Number analyzed (Participants) | 177 | 172 | 349
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.6) | 45.6 (11.3) | 45.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 117 | 255
  Male | 39 | 55 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 168 | 162 | 330
  Unknown or Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 18 | 32
  White | 155 | 149 | 304
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Montgomery Åsberg Depression Rating Scale (MADRS)
Description: Mean change from Week 8 (baseline) to Week 14 in MADRS total score, a 10-item, ordinal rating scale (0=no symptoms; 60=most severe symptoms). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (Week 8) and Week 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 174 | 169
units on a scale | -10.12 (0.74) | -6.39 (0.74)
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; The sample size for the study was based on the primary outcome measure. The study was powered at 90% to detect a treatment difference between adjunctive aripiprazole and adjunctive placebo of 3.75, assuming a standard deviation of 10.5 and a two-sided alpha level of 0.05. The null-hypothesis was the lack of a treatment difference; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -3.73, 95% CI [-5.44 to -2.02]

2. Secondary Outcome: Mean Change in Sheehan Disability Scale (SDS) Mean Score
Description: Mean change from Week 8 (baseline) to Week 14 in SDS Mean Score, a 3-item, ordinal scale (0=unimpaired; 30=highly impaired). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (Week 8) and Week 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 160 | 160
units on a scale | -1.22 (0.21) | -0.80 (0.20)
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; To protect the overall (primary and key secondary efficacy analysis) alpha level of 0.05, for this key secondary endpoint a hierarchical testing procedure was followed such that formal testing would take place conditional on the primary efficacy analysis showing a statistically significant difference; Test type: Superiority or Other; p = 0.075, t-test, 2 sided; Mean Difference (Final Values) = -0.42, 95% CI [-0.88 to 0.04]

3. Secondary Outcome: Mean Change in SDS Item Score (Social Life)
Description: Mean change from Week 8 (baseline) to Week 14 in SDS Social Life Item Score, 1 item from a 3-item, ordinal scale (0=unimpaired; 10=highly impaired). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (Week 8) and Week 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 160 | 160
units on a scale | -1.18 (0.24) | -0.65 (0.23)
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p = 0.052, t-test, 2 sided — No adjustment for multiple comparisons was implemented for this secondary endpoint; Mean Difference (Final Values) = -0.53, 95% CI [-1.06 to 0.00]

4. Secondary Outcome: Mean Change in SDS Item Score (Family Life)
Description: Mean change from Week 8 (Baseline) to Week 14 in SDS Family Life Item Score, 1 item from a 3-item, ordinal scale (0=unimpaired; 10=highly impaired). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (Week 8) and Week 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 160 | 160
units on a scale | -1.39 (0.24) | -0.82 (0.23)
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p = 0.037, t-test, 2 sided — No adjustment for multiple comparisons was implemented for this secondary endpoint; Mean Difference (Final Values) = -0.57, 95% CI [-1.10 to -0.03]

5. Secondary Outcome: Mean Change in SDS Item Score (Work/School)
Description: Mean change from Week 8 (baseline) to Week 14 in SDS Work/School Item Score, 1 item from a 3-item, ordinal scale (0=unimpaired; 10=highly impaired). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (Week 8) and Week 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 115 | 126
units on a scale | -0.75 (0.28) | -0.67 (0.26)
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p = 0.792, t-test, 2 sided — No adjustment for multiple comparisons was implemented for this secondary endpoint; Mean Difference (Final Values) = -0.08, 95% CI [-0.67 to 0.51]

6. Other Pre Specified Outcome: MADRS Response
Description: Number of subjects with a ≥50 percent reduction from Week 8 (baseline) in MADRS Total Score, a 10-item, ordinal rating scale to assess the severity of depressive symptoms (0=no symptoms; 60=most severe symptoms).
Time Frame: Baseline (Week 8) and Week 14
Measure: Number; unit: participants
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 174 | 169
participants
  Responders | 81 | 45
  Nonresponders | 93 | 124
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p < 0.001, CMH General Association Test — No adjustment for multiple comparisons was implemented for this secondary endpoint; Ratio of response = 1.74, 95% CI [1.31 to 2.32] — aripiprazole/placebo

7. Other Pre Specified Outcome: Clinical Global Impression (CGI)-Improvement Response
Description: Number of subjects with response relative to Week 8 (baseline). Response defined as score of 1 (very much improved) or 2 (much improved) on a 7-point, ordinal scale (1=very much improved; 7=very much worse).
Time Frame: Baseline (Week 8) and Week 14
Measure: Number; unit: Participants
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 174 | 169
Participants
  Responders | 109 | 74
  Nonresponders | 65 | 95
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiple comparisons was implemented for this secondary endpoint; Ratio of response = 1.43, 95% CI [1.17 to 1.74] — aripiprazole/placebo

8. Other Pre Specified Outcome: MADRS Remission
Description: Number of subjects in remission. Remission defined as as MADRS Total Score of <10 at 14 weeks, and a reduction of ≥50 percent from Week 8 (baseline) in MADRS, a 10-item, ordinal rating scale (0=no symptoms; 60=most severe symptoms).
Time Frame: Baseline (Week 8) and Week 14
Measure: Number; unit: participants
Arm/Group | Aripiprazole + ADT | Placebo + ADT
Number analyzed (Participants) | 174 | 169
participants
  Remission | 64 | 32
  No remission | 110 | 137
Statistical Analysis 1: Comparison: Aripiprazole + ADT vs Placebo + ADT; Test type: Superiority or Other; p < 0.001, CMH General Association Test — No adjustment for multiple comparisons was implemented for this secondary endpoint; Ratio of remission = 1.95, 95% CI [1.36 to 2.80] — aripiprazole/placebo

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 1/176 | 1/172
Other Adverse Events (participants affected / at risk) | 107/176 | 62/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=176) | Placebo (N=172)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=176) | Placebo (N=172)
VISION BLURRED (Eye disorders) | 13 | 3
INSOMNIA (Psychiatric disorders) | 15 | 9
RESTLESSNESS (Psychiatric disorders) | 22 | 6
HEADACHE (Nervous system disorders) | 15 | 14
AKATHISIA (Nervous system disorders) | 32 | 6
DIZZINESS (Nervous system disorders) | 9 | 5
SOMNOLENCE (Nervous system disorders) | 10 | 1
NAUSEA (Gastrointestinal disorders) | 7 | 10
DIARRHOEA (Gastrointestinal disorders) | 10 | 13
CONSTIPATION (Gastrointestinal disorders) | 10 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 13
FATIGUE (General disorders) | 16 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.